CLINICAL TRIAL: NCT00455000
Title: A Phase I, Randomized, Placebo Controlled, Double Blind Dose Escalation Study Of The Safety, Tolerability, Pharmacokinetics,Pharmacodynamics, And Immunogenicity Of A Single Intravenous Dose Of PF-04360365 In Adults With Mild To Moderate Alzheimer's Disease
Brief Title: A Phase I, Single IV Dose Of PF-04360365 In Adults With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9951001
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment (Experimental): 5 possible active doses
  Interventions: Biological: PF-04360365
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PF-04360365 — Monoclonal antibody
  Arms: Active treatment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is determine whether a single IV dose of PF-04360365 is safe and well tolerated in Adults with Mild to Moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or Females of non-childbearing potential, age 50-85
* Diagnosis of probable Alzheimer's disease, consistent with criteria from both: 1) National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA); and 2)Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* Mini-mental status exam score of 16-26 inclusive
* Rosen-Modified Hachinski Ischemia Score < or = 4

Exclusion Criteria:

* Diagnosis or history of other dementia or neurodegenerative disorders
* Diagnosis or history of clinically significant cerebrovascular disease
* Specific findings on magnetic resonance imaging (MRI): cortical infarct, micro hemorrhage, multiple white matter lacunes, extensive white matter abnormalities
* History of autoimmune disorders
* History of allergic or anaphylactic reactions

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To examine the safety, tolerability, and pharmacokinetics of a single dose of PF-04360365 in subjects with mild to moderate AD for one year following dosing. | 366 days

SECONDARY OUTCOMES:
To characterize the pharmacokinetic, pharmacodynamic and immunogenicity profile of PF-04360365 for one year following dosing. | 366 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Australia (3):
  - Pfizer Investigational Site, Heidelberg West, Victoria
  - Pfizer Investigational Site, Fremantle, Western Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Canada (3):
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Stockholm, Sweden
- Pfizer Investigational Site, Southampton, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951001&StudyName=A%20Phase%20I%2C%20Single%20IV%20Dose%20Of%20PF-04360365%20In%20Adults%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease